CLINICAL TRIAL: NCT02882763
Title: Zurich Equity Prevention Project Parental Participation and Integration
Brief Title: Early Support From Birth Onwards: ZEPPELIN
Acronym: ZEPPELIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Applied Sciences of Special Needs Education (Other)
Collaborators: Swiss National Science Foundation (Other); Jacobs Foundation (Unknown); Stiftung Mercator Schweiz (Unknown); Ernst Göhner Stiftung (Unknown); Paul Schiller Stiftung (Unknown); Vontobel-Stiftung (Unknown); Lotteriefonds des Kantons Zürich (Unknown); Bundesamt für Migration (BFM) (Unknown); Schweizerische UNESCO-Kommission (Unknown); University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ZEP_0-3_FU
Record Dates: First submitted 2016-07-28; First posted 2016-08-30 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Early Intervention (Education)
Keywords: Early intervention; ECCE; Intervention study; Child development; At-risk families; Psychosocial stress; Prevention; Educational opportunities; Randomized controlled trial; Evaluation; Parenting; Parent-child interaction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Parents As Teachers (PAT) (Experimental): c.f. intervention
  Interventions: Other: Parents As Teachers (PAT)
- control group condition (No Intervention): Families in the control group condition did not receive the home visiting program PAT, but were informed about support services in their community. The use of these services was permitted for ethical reasons; however, parents were regularly asked about the nature and intensity of the retrieved services. Additionally, all parents received incentives, such as greeting cards, small birthday presents, and monetary reimbursements.

INTERVENTIONS:
Other: Parents As Teachers (PAT) — A trained PAT parent educator (pediatric nurses in this study) visits families at their homes, approximately two times a month (individual frequencies may vary depending on specific risk factors) until the children are three years old. PAT is an educational home visitation program that aims to a) help parents to understand child developmental aspects and improve their parenting skills, b) detect developmental shortcomings, c) prevent child abuse and neglect, and d) enhance school preparedness. Additionally, the project offers monthly group meetings.
  Arms: Parents As Teachers (PAT)

SUMMARY:
ZEPPELIN (Zurich Equity Prevention Project with Parents Participation and Integration) is a longitudinal, randomized controlled intervention study. The main objective is to examine the effectiveness of the early intervention program "Parents As Teachers" (PAT) in psychosocially disadvantaged families. This includes four aims:

1. Identification of children at risk at an early age, using an interdisciplinary network;
2. Investigation of the acceptability of the program by the parents;
3. Evaluation of the intervention process and efficacy during and immediately after program implementation;
4. Evaluation of the efficacy in terms of child academic performance.

DETAILED DESCRIPTION:
The preschool years represent a critical time period, with major developmental milestones in cognitive, linguistic, motoric, and emotional areas. Families tend to manage this sensitive phase in different ways, which results in an uneven distribution of educational opportunities at school entry. However, prior evidence shows that these disparities can be reduced by means of evidence-based programs in early childhood care and education (ECCE). The main focus is on the prevention of learning and behavioral disorders; for small children, this occurs by means of strengthening parenting skills.

ZEPPELIN (Zurich Equity Prevention Project with Parents Participation and Integration) is a longitudinal, randomized controlled intervention study. The main objective is to examine the of the early intervention program "Parents As Teachers" (PAT) in psychosocially disadvantaged families. This includes four aims:

1. Identification of children at risk at an early age, using an interdisciplinary network;
2. Investigation of the acceptability of the program in parents;
3. Evaluation of the intervention process and efficacy during and immediately after program implementation;
4. Evaluation of the efficacy in terms of child academic performance.

Families were recruited in the suburbs of Zurich, Switzerland, shortly before or after giving birth. Baseline measurements were conducted at 3 months postnatal (t0), before participants were assigned to either the intervention group (IG, receiving the early intervention program PAT) or control group (CG) condition, using a stratified block randomization. Follow-up data was collected at three measurement time points around the first, second and third birthday of the children (t1, t2, t3).

Further follow-up measurements will be conducted in 2017 (t4; in the 1st year of kindergarten), 2018 (t5; in the 2nd year of kindergarten), 2019 (t6; after school transition), and in 2021 (t7; in the 3rd year of primary school). This will allow us to investigate medium-term and long-term effects of early developmental conditions.

ZEPPELIN 0-3 is the first ECCE program in Switzerland that specifically targets and recruits at risk families from birth on. Families then participate in an experimental field study including a longitudinal control group comparison. As such, ZEPPELIN fills an important gap in the current literature.

ELIGIBILITY:
Inclusion Criteria:

* Families shortly before or after child birth
* At risk situations (presence of at least two items from the core fields described below, while protective factors attenuating these risks appear absent)

Risk factors: core fields

* Personal risks, such as neglected appearance (subjective rating based on visual impression), low level of education (no further education after compulsory school years), early parenthood (mother younger than 20 years), alcohol and drug abuse, illness, disability, violence, unwanted pregnancy
* Familial risks, such as lack of self-management and planning skills), single parents, siblings with an age difference of 18 months or less, serious partnership conflicts (close to break up)
* Social risks, such as lack of social integration and support (no or only very few relationships outside the family), antisocial environment (violence, crime, prostitution)
* Material risks, such as confined living space (less than one room per person), unemployment (one or both parents), financial problems (dependency on welfare, debts)

Exclusion Criteria:

* Factors that may mitigate the risks, such as familial support, stable and reliable parents, clear and transparent family structures
* Immigrants without a permanent residence permit
* Severe illness or disability of the child or of the parents which require hospitalization or long-term treatment
* Other ongoing intensive treatments or child protection procedures

Max Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 213 (Actual)
Dates: Start 2011-09; Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Child development assessed with the Bayley Scale of Infant and Toddler Development (BSID III) | up to 3 years
  Bayley Scale of Infant and Toddler Development (BSID III)
Child development assessed with the Snijders-Oomen nonverbal intelligence test (SON-R) | up to 7 years
  Snijders-Oomen nonverbal intelligence test (SON-R)
Child development assessed with the Developmental Observation Scales (EBD 48-72) | up to 1 year
  German Developmental Observation Scales for child care centers (EBD 48-72)
Language skills assessed with the Language Evaluation Short form SBE-2-KT; SBE-3-KT) | up to 3 years
  Language evaluation short form (SBE-2-KT; SBE-3-KT)
Mathematical skills assessed with the TEDI-MATH test | up to 5 years
  Mathematical skills (TEDI-MATH)
Language skills assessed with the German test "Linguistically Competent" | up to 5 years
  "Linguistically Competent"
Child Health assessed with the Health questionnaire | up to 9 years
  Health questionnaire
Child Behavior assessed with the Child Behaviour Checklist (CBCL) | up to 6 years
  Child Behaviour Checklist (CBCL)
Child Behavior assessed with the Strengths and Difficulties Questionnaire (SDQ) | up to 5 years
  Strengths and Difficulties Questionnaire (SDQ)
Parent-child interaction assessed with the Child-Adult-Relationship-Experimental Index (CARE-Index) | up to 4 years
  Child-Adult-Relationship-Experimental Index (CARE-Index)
Parent-child interaction assessed with the Emotional Availability (EA) Scales | up to 3 years
  Emotional Availability (EA) Scales
Home environment assessed with the Home Observation Measurement of the Environment (HOME) | up to 7 years
  Home Observation Measurement of the Environment (HOME)

SECONDARY OUTCOMES:
Risk and protective factors assessed with the Heidelberg Stress Scale (HBS) | up to 8 years
  Heidelberg Stress Scale (HBS)
Risk and protective factors assessed with the German version of the Parenting-Stress-Index (EBI) | up to 3 years
  German version of the Parenting-Stress-Index (EBI)
Social network assessed with the Social Network Scales | up to 10 years
  Social Network Scales
Parental self-efficacy assessed with the Self-Efficacy in Infant Care Scale (SICS) | up to 4 years
  Self-Efficacy in Infant Care Scale (SICS)
Parental self-efficacy assessed with the Parenting Sense of Competence Scale (PSOC) | up to 3 years
  Parenting Sense of Competence Scale (PSOC)
Parental depressivity assessed with the subscale of the Brief Symptom Inventory (BSI) | up to 6 years
  Depressive symptoms (subscale BSI)
Educational attitudes assessed with the German test Educational Attitudes Scale (EMKK) | up to 4 years
  German "Educational Attitudes Scale" (EMKK)
Parenting assessed with the Alabama Parenting Questionnaire (APQ) | up to 3 years
  Alabama Parenting Questionnaire (APQ)

OTHER OUTCOMES:
Chronic biological stress assessed with nail cortisol concentrations (NCC) | up to 6 years
  Nail cortisol concentrations (NCC)
Chronic biological stress assessed with methylation in the FK506 binding protein 5 (FKBP5) gene | up to 6 years
  Methylation in the FK506 binding protein 5 (FKBP5) gene
Self-control assessed with the Watch-and-Wait Task | up to 7 years
  Watch-and-Wait Task
Dental health assessed with a Dental examination | up to 6 years
  Dental examination
Chronic biological stress assessed with methylation in the nuclear receptor subfamily 3 group C member 1 (NR3C1) gene | up to 6 years
  methylation in the nuclear receptor subfamily 3 group C member 1 (NR3C1) gene

CONTACTS AND LOCATIONS:
Overall Officials: Alex Neuhauser, lic. phil., Principal Investigator — University of Applied Sciences of Special Needs Education; Andrea Lanfranchi, Prof. Dr., Study Chair — University of Applied Sciences of Special Needs Education
Locations (1):
- University of Applied Sciences of Special Needs Education, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
After summer 2017 at the Swiss Centre of Expertise in the Social Sciences (FORS)

REFERENCES:
- [Background] Lanfranchi A, Neuhauser A. ZEPPELIN 0-3: Theoretische Grundlagen, Konzept und Implementation des frühkindlichen Förderprogramms "PAT -Mit Eltern Lernen". Frühe Bildung 2(1): 3-11, 2013.
- [Background] Neuhauser, A. A closer look at the effectiveness of early childhood education in at-risk families. Mental Health and Prevention 2(3-4): 43-57, 2014.
- [Background] Lanfranchi A, Neuhauser A. ZEPPELIN 0-3 - Förderung ab Geburt mit "PAT - Mit Eltern lernen". Sonderpädagogische Förderung heute, 56 (4): 437 - 442, 2011.
- [Background] Lanfranchi A, Sindbert R. Das Förderprogramm PAT-Mit Eltern Lernen - Eltern-Kind-Konzepte auf den Punkt gebracht. Frühförderung interdisziplinär, 32(2), 108-112, 2013.
- [Background] Templer F, Lanfranchi A, Neuhauser A. ZEPPELIN 0-3: Frühe Förderung ab Geburt mit dem Programm
- [Background] Lanfranchi A. Frühkindliche selektive Prävention bei Kindern aus Familien in Risikosituationen - Stigmatisierungsgefahren und Entwicklungschancen. Familiendynamik, 39(3), 188-199, 2014.
- [Background] Lanfranchi A, Sempert W. Wirkung frühkindlicher Betreuung auf den Schulerfolg Follow-up der Nationalfonds-Studie "Schulerfolg von Migrationskindern". Bern: Edition SZH, 2012.
- [Background] Lanfranchi A. Familienergänzende Betreuung. In M. Stamm & D. Edelmann (Eds.), Frühkindliche Bildung, Betreuung und Erziehung: Was kann die Schweiz lernen? (S. 97-121). Bern: Haupt, 2010.
- [Background] Lanfranchi A, Burgener Woeffray A. Familien in Risikosituationen durch frühkindliche Bildung erreichen. In M. Stamm & D. Edelmann (Eds.), Handbuch Frühkindliche Bildungsforschung (S. 603-616). Wiesbaden: VS/ Springer, 2013.
- [Result] Neuhauser A, Ramseier E, Schaub S, Burkhardt SCA, Templer F, Lanfranchi A. Hard to reach families - a methodological approach for early detection, recruitment, and randomization in an intervention study. Mental Health and Prevention, 3, 79-88, 2015.
- [Result] Neuhauser A. Predictors of maternal sensitivity in at-risk families. Early Child Development and Care (in press), 2016.